CLINICAL TRIAL: NCT01530880
Title: Aggressive Fever Control With Intravenous Ibuprofen After Non-traumatic Brain Hemorrhage
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: PI no longer at institution
Sponsor: Columbia University (Other)
Collaborators: Cumberland Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AAAI1788
Record Dates: First submitted 2012-02-08; First posted 2012-02-10 (Estimated); Results first posted 2017-08-28 (Actual); Last update posted 2017-08-28 (Actual); Status verified 2017-08

CONDITIONS: Fever
Keywords: Fever reduction; Fever burden; intravenous ibuprofen
MeSH Terms: conditions — Fever | interventions — Ibuprofen; Acetaminophen; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intravenous Ibuprofen (Experimental): Patients assigned to the ibuprofen treatment group will receive a 400 mg IV ibuprofen bolus over 30 minutes followed by an infusion of ibuprofen at 85 mg/hr.
  Interventions: Drug: Intravenous Ibuprofen
- Standard of Care (Other): Patients assigned to the standard of care group will be given 650 mg of oral acetaminophen and continue to receive 650 mg of oral acetaminophen every 6 hours as needed to maintain temperature < 38.3 C (100.9 F).
  Interventions: Drug: Acetaminophen (Standard of Care)

INTERVENTIONS:
Drug: Intravenous Ibuprofen — Ibuprofen 400 mg/100 mL intravenous (IV) over 30 minutes, followed by a continuous infusion of 2000 mg/500 mL at 85 mg/hour (21 mL/hour) for up to post bleed day 14 or discharge from the Neuro ICU, whichever comes first
  Other Names: Caldolor
  Arms: Intravenous Ibuprofen
Drug: Acetaminophen (Standard of Care) — Acetaminophen 650 mg via oral/nasogastric tube every 6 hours as needed for T>=38.3 C (100.9 F) for up to post bleed day 14 or discharge from the Neuro ICU, whichever comes first.
  Other Names: Tylenol
  Arms: Standard of Care

SUMMARY:
Fever, defined as temperature higher than 38.3C (100.9 F), is common in patients with head injuries and is associated with poor recovery after injury. The current standard of care is to use oral acetaminophen (Tylenol) followed by a body cooling device. This method can effectively reduce fever but results in a high rate of shivering. Shivering is stressful to the heart and can further worsen brain injury. Methods to combat shivering have been developed and are successful in limiting the stress in the majority of patients that use a body cooling device. However, the drugs used to control shivering are sedating and may also interfere with brain recovery.

The purpose of this study is to assess whether ibuprofen given intravenously is more effective in combating fever than the current standard of care. Should results from this study demonstrate that ibuprofen infusion is effective, a larger study will be conducted to determine whether this aggressive fever control regimen leads to improved recovery after brain injury.

DETAILED DESCRIPTION:
This is an open-label, investigator initiated single center, randomized, prospective study. Subjects meeting enrollment criteria will be randomly assigned 1:1 to one of two groups:

1. Standard Care: Acetaminophen 650 mg via oral/nasogastric tube every 6 hours as needed for T>=38.3 C (100.9 F) for up to post bleed day 14 or discharge from the Neuro ICU, whichever comes first.
2. Ibuprofen 400 mg/100 mL NS IV over 30 minutes, followed by a continuous infusion of 2000 mg/500 mL NS at 85 mg/hour (21 mL/hour) for up to post bleed day 14 or discharge from the Neuro ICU, whichever comes first.

Patients/surrogates will be approached for consent and randomized upon admission. Therapy will only be initiated once a patient becomes febrile (>=38.3 C, 100.9 F). The use of temperature modulating devices will be permitted as per institutionally approved guidelines in those patients continuing to demonstrate a fever (T>38.3 C, 100.9 F) with either therapy.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Aneurysmal subarachnoid hemorrhage (SAH), Hunt Hess grade >= 3, 24 hours after admission.
* Intracerebral hemorrhage (ICH), Glasgow Coma Scale (GCS) < 10
* Presence of intraventricular hemorrhage on initial brain computerized tomography (CT) scan

Exclusion Criteria:

* Imminent death within 72 hours of admission.
* Plan for discharge from the Neuro intensive care unit (ICU) within 72 hours of admission.
* Diagnosis with sepsis (Systemic inflammatory response syndrome (SIRS) criteria plus the presence of known or suspected infection)
* Presence of coagulopathy (international normalized ratio (INR) > 1.7)
* Thrombocytopenia (platelet count < 100,000)
* History of gastrointestinal bleed
* Abnormal liver function tests (aspartate aminotransferase (AST)/alanine aminotransferase (ALT)/alkaline phosphatase (AP)/Gamma-glutamyl transferase (GGT) 2x normal)
* Hypersensitivity to ibuprofen
* Pregnancy as determined by urine beta human chorionic gonadotropin (hCG), or lactating postpartum women
* Renal impairment (Creatinine > 1.5 mg/dL)
* Measured body weight < 50 kg

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2012-10; Primary Completion 2016-03-17 (Actual); Study Completion 2016-03-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: J. Michael Schmidt, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Medical Center, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- All Subjects: Includes subjects from both arms as this information is only available for all subjects and not per arm.
Period: Overall Study
Arm/Group | All Subjects
Started | 35
Completed | 35
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Includes subjects from both arms as this information is only available for all subjects and not per arm.
Groups:
- All Subjects: Includes subjects from both arms.
Arm/Group | All Subjects
Number analyzed (Participants) | 35
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 29
  >=65 years | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30
  Male | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 19
  Not Hispanic or Latino | 16
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Prevalence of Fever Burden
Description: Reduction in fever burden (degrees C x hours) with intravenous ibuprofen infusion as compared to oral acetaminophen over duration of treatment. Fever burden is calculated hourly by subtracting each patient's recorded temperature (from either a bladder or esophageal temperature probe) from 37 degrees C.
Time Frame: Up to14 days
Population: PI left before data could be analyzed and data collection was incomplete.
Arm/Group | Intravenous Ibuprofen | Standard of Care
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Mean Difference in Inflammatory Markers
Description: Mean difference in markers of inflammation between IV ibuprofen and standard of care groups
Time Frame: Up to 14 days
Population: PI left before data could be analyzed and data collection was incomplete.
Arm/Group | Intravenous Ibuprofen | Standard of Care
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Difference in Cost Between Ibuprofen and Acetaminophen
Description: Cost analysis of aggressive fever control (AFC) between patients randomized to either intravenous ibuprofen infusion or standard of care (oral acetaminophen).
Time Frame: Up to 14 days
Population: PI left before data could be analyzed and data collection was incomplete.
Arm/Group | Intravenous Ibuprofen | Standard of Care
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Bleeding Incidence
Description: Incidence of bleeding (defined by a priori criteria)
Time Frame: Up to 14 days
Population: PI left before data could be analyzed and data collection was incomplete.
Arm/Group | Intravenous Ibuprofen | Standard of Care
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | All Subjects
All-Cause Mortality (participants affected / at risk) | 0/35
Serious Adverse Events (participants affected / at risk) | 0/35
Other Adverse Events (participants affected / at risk) | 0/35

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes